CLINICAL TRIAL: NCT06165549
Title: A Randomized Controlled Double-Blind Trial of Light Therapy for Internet Gaming Disorder
Brief Title: Light Therapy for Internet Gaming Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinan University Guangzhou (Other)
Responsible Party: Principal Investigator, Qian Tao, Professor Tao, Jinan University Guangzhou
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Internet Gaming Disorder
Record Dates: First submitted 2023-11-27; First posted 2023-12-11 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Internet Gaming Disorder; Light Therapy
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Light therapy (Experimental): about 30 individuals with internet gaming disorder will be randomly assigned to the light therapy group
  Interventions: Other: Light therapy
- Light placebo (Placebo Comparator): about 30 individuals with internet gaming disorder will be randomly assigned to the light placebo group
  Interventions: Other: Light placebo therapy
- EABM training group (Other): about 30 individuals with internet gaming disorder will be randomly assigned to the EABM training group
  Interventions: Other: Emotion Bias Modification Training

INTERVENTIONS:
Other: Light therapy — The light therapy will be administered by custom-made light boxes (LED) with adjustable brightness. The light intensity will be set at 5000 Lux. The intervention will consist of daily exposure for 30 minutes in the morning. The whole intervention includes 14 days.
  Arms: Light therapy
Other: Light placebo therapy — The light placebo intervention will be administered by custom-made light boxes (LED) with adjustable brightness. The light intensity will be set at less than 200 Lux. The intervention will consist of daily exposure for 30 minutes in the morning. The whole intervention includes 14 days.
  Arms: Light placebo
Other: Emotion Bias Modification Training — The training aims at associating gaming pictures with negative words and pictures of healthy activities with positive words. Gaming pictures are always presented with a pair of negative words. Pictures of healthy activities are always presented with a pair of positive words. Each picture is presented with a fixed pair of words. Participants will be instructed to select one word to get the most monetary reward. Specifically, selecting a fixed word of the word-pair will be associated with a high probability (eighty percent) of getting a monetary reward and a low probability (twenty percent) of no reward, and probabilities will be reversed for the other word. Each training run will comprise 100 gaming picture trials and 100 healthy-activity picture trials, presented in a pseudo-randomized order. Participants will receive two training runs every day. The whole training includes 14 days.
  Arms: EABM training group

SUMMARY:
This project aims to investigate (1) the efficacy of light therapy on internet gaming disorder (IGD); (2) the underlying neural mechanisms of such efficacy

ELIGIBILITY:
Inclusion Criteria:

1. the 5th edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-5 ) recommended diagnosis of Internet gaming disorder;
2. the scores of the Young-Internet addiction Test ≥ 50;
3. playing internet games ≥15 h/week for ≥1 year

Exclusion Criteria:

1. current or history of psychiatric or neurological illness;
2. current or history of use of illegal substances and other addictions;
3. current use of psychotropic medications ;
4. any history of head trauma, presence of metal in the body or other contraindication to functional MRI scanning;
5. photosensitivity disorders, such as systemic lupus erythematosus and chronic actinic dermatitis.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2023-12-16 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
changes in IGD severity | baseline , within one day after intervention, and 4-week after intervention
  The scores of IGD severity will be assessed with the internet addiction test for internet gaming disorder.
changes in weekly gaming time | baseline and within 1 day after intervention
  weekly gaming time will be recorded by Software.
changes in withdrawal symptoms | baseline and within 1 day after intervention
  The scores of withdrawal symptoms will be assessed with the mood and physical symptoms scale.
change of BOLD signals | baseline and within 1 day after intervention
  Task-based fMRI and resting state fMRI.
changes in craving | baseline and within 1 day after intervention
  Craving will be assessed using a Visual Analog Scale during a cue-reactivity task.

SECONDARY OUTCOMES:
changes in gaming-related compulsive behaviors | baseline and within 1 day after intervention
  The scores of gaming-related compulsive behaviors will be assessed with the Yale-Brown Obsessive-Compulsive Scale modified for internet gaming disorder.
changes in gaming-related compulsive thoughts | baseline and within 1 day after intervention
  The scores of gaming-related compulsive thoughts will be assessed with the Yale-Brown Obsessive-Compulsive Scale modified for internet gaming disorder.
changes in the quality and patterns of sleep | baseline and within 1 day after intervention
  The scores of the quality and patterns of sleep will be assessed with the Pittsburgh Sleep Quality Index (PSQI).
changes in the severity of depression | baseline and within 1 day after intervention
  The scores of the severity of depression will be assessed with the Beck Depression Inventory（BDI）
changes in the severity of anxiety | baseline and within 1 day after intervention
  The scores of the severity of anxiety will be assessed with the Beck Anxiety Inventory (BAI)
changes in the severity of two emotion regulation strategies, cognitive reappraisal and expressive suppression | baseline and within 1 day after intervention
  The scores of emotion regulation strategies will be assessed with the Emotion Regulation Questionnaire (ERQ)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - South China Normal University, Guangzhou, Guangdong
  - Jinan University, Guangdong, Guangzhou